CLINICAL TRIAL: NCT03415360
Title: Percutaneous Cryoablation in the Treatment of Neuropathic Pain Post Limb Amputation
Brief Title: Cryolesion in Treatment of Phantom Limb Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Dariusz Tomaszewski, Adjunct professor, Military Institute od Medicine National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 681006-6
Record Dates: First submitted 2018-01-13; First posted 2018-01-30 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Phantom Limb Pain; Stump Neuralgia; Pain, Phantom
Keywords: cryoablation
MeSH Terms: conditions — Phantom Limb; Neuralgia | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cryoablation (Other): peripheral nerve cryoablation
  Interventions: Procedure: cryoablation

INTERVENTIONS:
Procedure: cryoablation — cryoablation of nerve responsible for phantom limb pain

SUMMARY:
Assessment of pain intensity on the NRS. Assessment of the quality of life by SF-36 and AIS. Diagnostic/prognostic nerve block with 5 ml of 2% lidocaine under real-time ultrasound control with confirmation of the correct position of the needle using a peripheral nerve stimulator.

Reassessment of pain intensity on the NRS 30 minutes after local anesthetic block.

Cryoablation under real-time ultrasound control if the NRS value is reduced by ≥ 2 points.

If pain intensity on the NRS reduced by less than 2 points, reassessment 60 minutes after local anesthetic block.

Cryoablation under real-time ultrasound control if the NRS value is reduced by ≥ 2 points.

If pain intensity on the NRS reduces by less than 2 points 60 minutes after local anesthetic block cryoablation will not be performed.

Cryoablation effect will be evaluated 24 hours, 7 days, 30 days, 3 months, 6 months post procedure.

* 24 hours after the procedure - assessment of pain intensity and quality of life
* 7 days after the procedure - assessment of pain intensity
* 30 days after the procedure - assessment of pain intensity and quality of life
* 3 months after the procedure - assessment of pain intensity
* 6 months after the procedure - assessment of pain intensity and quality of

ELIGIBILITY:
Inclusion Criteria:

* Status post amputation of a lower or upper limb
* Pain related to amputation as determined by referring physician and investigator
* Informed consent of patient to enter the study
* Reduction of pain after the diagnostic/prognostic anesthetic block of the relevant main peripheral nerves under ultrasonography guidance in an analogous fashion to the cryoablation procedure

Exclusion Criteria:

* Pregnancy
* Active infection in the area of the planned intervention
* Blood coagulation disorders
* Immunosuppression
* Significant spinal stenosis or spinal anomalies that result in differential nerve root pressures
* Significant disease or disorder that in the opinion of the Principal Investigator would preclude the safe performance of the anesthetic block or cryoablation
* Participation in another investigational trial involving systemic administration of agents of unknown chemical composition.
* No reduction of pain after the diagnostic block of the relevant main peripheral nerves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain | T1: before cryoablation; T2: 24 hours after cryoablation; T3: 7 days after cryoablation; T4: 30 days after cryoablation; T5: 3 months after cryoablation; T6: 6 months after cryoablation.
  Assessment of pain intensity pre- and post - cryoablation on the NRS (numeric rating scale).
  Numeric Rating Scale (NRS) is a unidimensional measure of pain intensity in adults. This is a 11-point numeric scale ranges from '0' (minimum, "no pain") to '10' (maximum, "pain as bad as one can imagine"). The lower the NRS value, the better clinical outcome.

SECONDARY OUTCOMES:
The quality of life (SF-36) | A1: before cryoablation; A2: 24 hours after cryoablation; A3: 30 days after cryoablation; A4: 6 months after cryoablation.
  Assessment of the quality of life pre- and post - cryoablation on SF-36. 36-Item Short Form Survey (SF-36) is a 36-item questionnaire which measures quality of life across eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health.
  For each of the eight domains that the SF36 measures an aggregate percentage score is produced. The percentage scores range from 0% (lowest or worst possible level of functioning) to 100% (highest or best possible level of functioning).
The quality of life (AIS) | A1: before cryoablation; A2: 24 hours after cryoablation; A3: 30 days after cryoablation; A4: 6 months after cryoablation.
  Assessment of the quality of life pre- and post - cryoablation on AIS. The Acceptance of Illness Scale (AIS) consists of eight statements describing negative impact of poor health status and its consequences for patients' functioning. The scoring for each statement varies from 1 (poor adaptation to the disease) to 5 (full acceptance of the disease). The total score ranges between 8 and 40. The lower score, the poorer acceptance of disease and more severe restrictions caused by condition. A high score means acceptance of patient's own health status and lack of negative emotions related to illness.

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Tomaszewski, Study Chair — Military Institute of Medicine
Locations (1):
- Military Institute of Medicine, Warsaw, Poland